CLINICAL TRIAL: NCT04490265
Title: Suicide Prevention for Patients With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Veterans BioMedical Research Institute (Other)
Collaborators: Rutgers University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5R56MH121555 (NIH)
Record Dates: First submitted 2020-07-06; First posted 2020-07-29 (Actual); Results first posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Suicide; Chronic Pain
MeSH Terms: conditions — Suicide; Chronic Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Problem-Solving Treatment (Experimental): Our PST is 12-weeks and teaches patients strategies to address real-life problems.20 Sessions are once a week for one hour except for the first session, which is two hours. The treatment has four main goals: 1. Safety planning; 2. Problem-orientation-addressing how patients approach problems; 3. Planful problem-solving or a logical approach to address problems; 4. Behavioral activation of daily activities. Patients are provided weekly worksheets on problem-solving and receive weekly assessment of emotional state and suicidal ideation monitoring.
  Interventions: Behavioral: Problem-solving treatment
- Supportive Psychotherapy (Placebo Comparator): Our control will be supportive psychotherapy which will focus on discussing weekly stressors in a supportive, non-directive way. Session content is patient-driven, and sessions focus on emphasizing the patients' strengths, following patients' emotional affect, and building a therapeutic alliance. Participants will be asked to generate the topic they would like to discuss for the session and will complete a worksheet between sessions noting emotional events throughout their week ("A time when I felt stressed was …" ) in order to help identify experiences for discussion in session. Participants will be informed that the control condition is supportive and non-directive, and that providers will not engage in problem-solving. Providers will be taught to use reflective listening, clarification, empathy, and validation. The control consists of 12 weekly sessions delivered via telephone or video.
  Interventions: Behavioral: Supportive Psychotherapy

INTERVENTIONS:
Behavioral: Problem-solving treatment — included in arm descriptions
  Arms: Problem-Solving Treatment
Behavioral: Supportive Psychotherapy — included in arm descriptions
  Arms: Supportive Psychotherapy

SUMMARY:
Patients with chronic pain and moderate suicide risk (n=60) will be randomized to receive remote-PST or remote-supportive psychotherapy. We will assess problem-solving deficits through self-report, objective neuropsychological assessment and caregiver report. We have used an adaptive design so that if there is strong evidence for target engagement, we will continue with the trial as a fully powered clinical trial (i.e., the end of the current proposal will act as the interim assessment) to the determine the efficacy of remote PST for patients with chronic pain and moderate suicide risk (n=190) to improve suicide outcomes.

DETAILED DESCRIPTION:
Every day, 120 people die from suicide, that is one person every 15 minutes.1 Suicide prevention treatments focus on those at highest risk and are primarily delivered as mental health treatments,2-5 and yet 70% of patients with suicide risk do not attend mental health treatment. Developing treatment for patients not served by existing suicide prevention programs will improve access to care and is necessary to stop suicide.

Patients with chronic pain in the US (100 million) have 2.6-times greater risk of suicide and those on long-term opioid treatment are at even greater risk. Unfortunately, they often do not receive mental health treatment and thus do not receive suicide prevention interventions. They do receive frequent healthcare for their pain providing an unmet opportunity to integrate suicide prevention into their treatment for pain.

Problem-solving treatment (PST) is an evidence-based approach that is available where patients want to receive treatment (e.g., primary care) and is efficacious for chronic pain. Importantly, PST targets problem-solving deficits which are known to increase risk of suicide, suggesting PST could be leveraged to reduce suicide risk. Deficits in problem-solving (an executive function of finding solutions to difficult issues) directly increase suicidal risk because they keep patients with active suicidal ideation from generating solutions to their problems (e.g., chronic pain), other than through suicide. Deficits in problem-solving also make it difficult to keep pain from impairing daily activities and social relationships. This indirectly increases suicide risk because impairment in daily activities increases feelings of burdensomeness and impairment in social relationships increases feelings of not belonging. Feelings of burdensomeness and of not belonging are key theoretical pathways to suicidal behavior.

Working with our clinical partners and patients, we developed a 12-week remote delivered PST for patients with chronic pain and moderate suicidal risk. The treatment addresses deficits in problem-solving by teaching patients strategies to address problems caused by chronic pain that increase risk of suicide (e.g., impairment in daily activities leading to feelings of burdensomeness). Our preliminary data suggests that PST is feasible, acceptable and may be efficacious. In a national survey we found 56% of patients with chronic pain and suicide risk were interested in problem-solving treatment. In a clinical pilot we were able to engage Veterans with chronic pain and suicide risk with 75% completing the treatment. Finally, in a clinical trial that randomized patients to 12 sessions of PST or 12 sessions of health education, we found that patients with chronic pain and moderate suicide risk (n=21) randomized to PST had a reduction in suicidal ideation and problem-solving deficits (self-report) as compared to health education.

The goal of the current proposal (R56) is to ensure PST is engaging problem-solving deficits. Patients with chronic pain and moderate suicide risk (n=60) will be randomized to receive remote-PST or remote-supportive psychotherapy. We will assess problem-solving deficits through self-report, objective neuropsychological assessment and caregiver report. We have used an adaptive design so that if there is strong evidence for target engagement, we will continue with the trial as a fully powered clinical trial (i.e., the end of the current proposal will act as the interim assessment) to the determine the efficacy of remote PST for patients with chronic pain and moderate suicide risk (n=190) to improve suicide outcomes.

Aim 1: Estimate the effect of remote-delivered PST on targets. We hypothesize that PST reduces our primary target, problem-solving deficits as assessed through (H1) self-report, (H2) objective neuropsychological assessment, (H3) caregiver report, as compared to supportive psychotherapy. We hypothesize that PST reduces our secondary targets (H1) feelings of burdensomeness and (H2) feelings of not belonging, as compared to supportive psychotherapy.

Exploratory Aim 2: Explore the effect size of PST as compared to supportive psychotherapy on suicide outcomes (intensity of suicidal ideation, difficulties coping with suicidal ideation) and chronic pain outcomes ((H4) chronic pain, (H5) pain related disability).

Our previous preliminary data suggests that PST is feasible, acceptable and may be efficacious. The goal of the current proposal (R56) is to confirm PST is engaging problem-solving deficits (measured through self-report and objective measures). Deliverable: At the end of the proposed trial, we will have the necessary information (in combination with our previous preliminary data) to inform a go/no-go decision on converting the current proposal into a fully powered clinical trial.

ELIGIBILITY:
Inclusion criteria will include:

* has a VA primary care provider and has had an in-person visit with a VA provider in the past year;
* pain that is (b1) musculoskeletal, defined as regional (joints, limbs, back, neck) or more generalized (chronic widespread pain);
* pain that is (b2) moderately severe, defined as a Brief Pain Inventory (BPI) intensity item score of 5 or higher for either "average" or "worst" pain in the past week;
* pain that is (b3) persistent, (i.e., ≥3 months)
* active suicidal ideation defined as scoring a 2 to 4 on the C-SSRS.

Exclusion Criteria:

* life-threatening condition
* severe cognitive impairment
* psychotic disorder
* pregnant or plans to become pregnant in the next year
* suicide attempt in the past year or hospitalization for suicide risk in the past year

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2023-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M McAndrew, PhD, Principal Investigator — VA NJHCS
Locations (1):
- VA NJHCS, East Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
If the subject agrees, their data will be submitted to the National Institute of Mental Health Data Archive (NDA) at the National Institutes of Health (NIH). NDA is a large database where deidentified study data from many National Institute of Mental Health (NIMH) studies is stored and managed.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Every 3 months data is uploaded
URL: https://nda.nih.gov

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrolled = Participants who enrolled into the study (n=60) Baseline = Participants who consented into the study and were randomized (n=44)
Period: Overall Study
Arm/Group | Problem-Solving Treatment | Supportive Psychotherapy
Started | 22 | 22
Completed | 19 | 16
Not Completed | 3 | 6

BASELINE CHARACTERISTICS:
Population: Baseline Analysis = participants who consented, were randomized, and completed baseline measures
Groups:
- Total: Total of all reporting groups
Arm/Group | Problem-Solving Treatment | Supportive Psychotherapy | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Continuous [Mean (Full Range); unit: years] | 48.2 [27 to 69] | 52.5 [32 to 75] | 50.4 [27 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 16 | 17 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 15 | 20 | 35
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 10 | 16 | 26
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 4 | 0 | 4
Social Problem-Solving [Mean (Standard Deviation); unit: units on a scale] | 82.16 (18.20) | 88.81 (22.33) | 85.65 (20.37)

OUTCOME MEASURES:

1. Primary Outcome: Social Problem-solving Inventory - Patient Report
Description: The Social problem-solving inventory - patient report measures problem-solving that is sensitive to change. In clinical research, the Social problem-solving inventory - patient report has been successfully used to elicit meaningful self-appraisals. The questionnaire is 52 items long. We will use the total score. Scores range from 0-100 with higher scores equaling better problem-solving.
Time Frame: Change from Baseline to 12 weeks
Population: Only individuals who provided data were analyzed.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Problem-Solving Treatment | Supportive Psychotherapy
Number analyzed (Participants) | 17 | 14
score on a scale | 8.12 [0 to 16.24] | 3.64 [-1.99 to 9.28]
Statistical Analysis 1: Comparison: Problem-Solving Treatment vs Supportive Psychotherapy; Test type: Superiority; Cohen's d = .33

2. Primary Outcome: Social Problem-solving Inventory - Patient Report
Description: The Social problem-solving inventory - patient report measures problem-solving that is sensitive to change. In clinical research, the Social problem-solving inventory - patient report has been successfully used to elicit meaningful self-appraisals. The questionnaire is 52 items long. We will use the total score.Scores range from 0-100 with higher scores equaling better problem-solving.
Time Frame: Change from Baseline to 6 months
Population: Only individuals who provided data were analyzed.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Problem-Solving Treatment | Supportive Psychotherapy
Number analyzed (Participants) | 13 | 17
score on a scale | 8.31 [0.91 to 15.70] | -.24 [-5.33 to 4.86]
Statistical Analysis 1: Comparison: Problem-Solving Treatment vs Supportive Psychotherapy; Test type: Superiority; Cohen's d = .78

3. Primary Outcome: Emotional Go No Go
Description: Emotional Go No Go measures attention and impulse inhibition. Inhibiting impulses is a key component of preventing impulsive behavior that can lead to suicide. Reported is the hit rate with scores from 0-1.0. Higher scores are better.
Time Frame: Change from Baseline to 12 weeks
Population: Only individuals who provided data were analyzed.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Problem-Solving Treatment | Supportive Psychotherapy
Number analyzed (Participants) | 12 | 7
score on a scale | -.01 [-.09 to .08] | .06 [-.03 to .15]

4. Primary Outcome: Means End Problem-Solving Task
Description: The Means End Problem-Solving Task consists of a series of scenarios, with each one identifying the beginning and end of a story. The subject's task is to come up with the middle of the story. Stories are scored according to how many steps to reaching the end the patient identifies. An increase in effective means generated is expected to drive reduction in suicide ideation. We report the total score, the range was 2-19. Scores higher=better problem-solving.
Time Frame: Change from Baseline to 12 weeks
Population: Only individuals who provided data were analyzed.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Problem-Solving Treatment | Supportive Psychotherapy
Number analyzed (Participants) | 14 | 17
score on a scale | -1.36 [-4.66 to 1.95] | 0.29 [-1.99 to 2.58]

5. Primary Outcome: Iowa Gambling Task
Description: The Iowa gambling task is a neuropsychological task of problem-solving. The participgoal of the task is to make money. Participants are presented four decks of cards and have to choose the best deck to make money. The Iowa gambling task has been shown to change after problem-solving therapy. Scores range from -100 to 100 with higher equaling better problem-solving.
Time Frame: Change from Baseline to 12-weeks
Population: Only individuals who provided data were analyzed.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Problem-Solving Treatment | Supportive Psychotherapy
Number analyzed (Participants) | 12 | 7
score on a scale | 23.33 [-3.77 to 50.44] | 26.14 [-27.73 to 80.01]

6. Primary Outcome: Emotional Stroop
Description: The emotional Stroop is a test of response inhibition. There are four category conditions: aggression, color, negative, and positive. Scores were derived based on the difference between the median latency of neutral condition subtracted from median latency of category conditions (unit=miliseconds) with higher scores equaling better problem-solving. Score range did not exceed -500 to 500.
Time Frame: Change from Baseline to 12 weeks
Population: Only individuals who provided data were analyzed.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Problem-Solving Treatment | Supportive Psychotherapy
Number analyzed (Participants) | 12 | 7
score on a scale
  Aggression | 59.21 [-24.19 to 142.60] | 13.50 [-52.15 to 79.15]
  Color | 123.00 [33.49 to 212.51] | 59.49 [-123.77 to 242.74]
  Negative | 55.50 [-77.95 to 188.95] | 72.71 [-101.21 to 246.64]
  Positive | 97.67 [22.15 to 173.18] | 71.14 [-80.86 to 223.15]

7. Secondary Outcome: Interpersonal Needs Questionnaire
Description: Feelings of burdensomeness and belongingness will be measured by the Interpersonal Needs Questionnaire (INQ). This measure is 18-item self-report questionnaire. The belonging subscale is 6 items and scores range from 6-42 with higher scores indicating less belonging, the burdensomeness subscale is 9 items and scores range from 9-63 with higher scores indicating greater burdensomeness.
Time Frame: Change from Baseline to 12 weeks, Baseline to 6 months
Population: Only individuals who provided data were analyzed.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Problem-Solving Treatment | Supportive Psychotherapy
Number analyzed (Participants) | 19 | 18
score on a scale
  Belonging - follow-up | -2.37 [-8.05 to 3.31] | -.81 [-6.54 to 4.91]
  Burden-follow-up | -4.37 [-7.44 to -1.29] | -.5 [-3.96 to 2.96]
  Belonging-6 months | -.4 [-5.26 to 4.46] | -.79 [-3.72 to 2.14]
  Burden - 6 months | -3.2 [-6.37 to -.03] | .11 [-4.22 to 4.43]
Statistical Analysis 1: Comparison: Problem-Solving Treatment vs Supportive Psychotherapy; Belonging Subscale change from baseline to 12-weeks; Test type: Superiority; Cohen's d = 0.14
Statistical Analysis 2: Comparison: Problem-Solving Treatment vs Supportive Psychotherapy; Belonging subscale Baseline to 6-months; Test type: Superiority; Cohen's D = 0.05
Statistical Analysis 3: Comparison: Problem-Solving Treatment vs Supportive Psychotherapy; Change in Burdensome subscale Baseline to 12-weeks; Test type: Superiority; Cohen's D = 0.60
Statistical Analysis 4: Comparison: Problem-Solving Treatment vs Supportive Psychotherapy; Change in Burdensome subscale Baseline to 6 months; Test type: Superiority; Cohen's D = 0.43

8. Other Pre Specified Outcome: Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: Columbia-Suicide Severity Rating Scale (C-SSRS) is the gold standard for suicide assessment and measures level and intensity of suicidal ideation, planning and preparation for suicidal behavior, and method and lethality of recent (past week) and past lifetime suicidal behavior. The intensity of ideation subscale (the summed score from five separate items on Part II; subscale range = 2-25) will be the primary dependent variable for the fully powered clinical trial. The intensity of ideation asks about the intensity of ideation in the past 6 months (e.g., the frequency, duration controllability). Higher scores are equal to greater ideation.
Time Frame: Change from Baseline to 12 weeks and Baseline to 6 months
Population: Only individuals who provided data were analyzed.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Problem-Solving Treatment | Supportive Psychotherapy
Number analyzed (Participants) | 11 | 14
score on a scale
  follow-up | -.82 [-3.38 to 1.75] | -1.14 [-4.08 to 1.79]
  6-months | -1.23 [-5.01 to 2.54] | -.5 [-3.43 to 2.43]
Statistical Analysis 1: Comparison: Problem-Solving Treatment vs Supportive Psychotherapy; Baseline to 12-weeks; Test type: Superiority; Cohen's D = 0.07
Statistical Analysis 2: Comparison: Problem-Solving Treatment vs Supportive Psychotherapy; Baseline to 6-months; Test type: Superiority; Cohen's D = 0.13

9. Other Pre Specified Outcome: Suicide Ideation Questionnaire (SIQ).
Description: Suicide Ideation Questionnaire (SIQ) is a 30-item self-report instrument designed to assess thoughts about suicide experienced during the prior month. This measure has strong internal consistency and construct validity. This measure will allow for supplementary investigation of ideation. Scores range from 7-210 with higher equaling worse ideation.
Time Frame: Change from Baseline to 12 weeks
Population: Only individuals who provided data were analyzed.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Problem-Solving Treatment | Supportive Psychotherapy
Number analyzed (Participants) | 18 | 16
score on a scale | -19.28 [-33.09 to -5.47] | -2.88 [-17.29 to 11.54]
Statistical Analysis 1: Comparison: Problem-Solving Treatment vs Supportive Psychotherapy; Test type: Superiority; Cohen's d = .60

10. Other Pre Specified Outcome: Suicide Ideation Questionnaire (SIQ).
Description: as for outcome 9
Time Frame: Change from Baseline to 6 months
Population: Only individuals who provided data were analyzed.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Problem-Solving Treatment | Supportive Psychotherapy
Number analyzed (Participants) | 14 | 18
score on a scale | -21.71 [-39.95 to -3.48] | -7.0 [-19.51 to 5.51]
Statistical Analysis 1: Comparison: Problem-Solving Treatment vs Supportive Psychotherapy; Test type: Superiority; Cohen's d = .52

11. Other Pre Specified Outcome: Suicide-Related Coping Scale
Description: The Suicide-Related Coping Scale captures an individual's perceived ability to use internal and external coping to problem-solve suicidal thoughts and urges. This measure was validated in a Veteran sample. The items in this measure capture the types of skills we expect Veterans to be able to use after learning problem-solving (i.e., "I recognize the circumstances that make me suicidal"). Scores range from 0-68 with higher scores indicating better coping.
Time Frame: Change from Baseline to 12 weeks
Population: Only individuals who provided data were analyzed.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Problem-Solving Treatment | Supportive Psychotherapy
Number analyzed (Participants) | 17 | 16
score on a scale | 1.94 [-2.76 to 6.64] | 4.06 [-1.63 to 9.75]
Statistical Analysis 1: Comparison: Problem-Solving Treatment vs Supportive Psychotherapy; Test type: Superiority; Cohen's d = .21

12. Other Pre Specified Outcome: Suicide-Related Coping Scale
Description: as for outcome 11
Time Frame: Change from Baseline to 6 months
Population: Only individuals who provided data were analyzed.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Problem-Solving Treatment | Supportive Psychotherapy
Number analyzed (Participants) | 15 | 18
score on a scale | 1.53 [-3.09 to 6.16] | 3.33 [-1.51 to 8.18]
Statistical Analysis 1: Comparison: Problem-Solving Treatment vs Supportive Psychotherapy; Test type: Superiority; Cohen's d = .20

13. Other Pre Specified Outcome: Pain Disability Index (PDI)
Description: Pain Disability Index (PDI) is a 7 item measure of the impact of pain on daily activities and social relationships. It will be used to assess disability from pain. The PDI ranges from 0-70 with higher scores indicating worse disability from pain.
Time Frame: Change from Baseline to 12 weeks
Population: Only individuals who provided data were analyzed.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Problem-Solving Treatment | Supportive Psychotherapy
Number analyzed (Participants) | 16 | 16
score on a scale | -4.88 [-9.88 to 0.13] | 2.13 [-4.13 to 8.38]
Statistical Analysis 1: Comparison: Problem-Solving Treatment vs Supportive Psychotherapy; Test type: Superiority; Cohen's d = 0.66

14. Other Pre Specified Outcome: Pain Disability Index (PDI)
Description: Pain Disability Index (PDI) is a 7 item measure of the impact of pain on daily activities and social relationships. It will be used to assess disability from pain.The PDI ranges from 0-70 with higher scores indicating worse disability from pain.
Time Frame: Change from Baseline to 6 months
Population: Only individuals who provided data were analyzed.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Problem-Solving Treatment | Supportive Psychotherapy
Number analyzed (Participants) | 14 | 18
score on a scale | -2.79 [-8.26 to 2.69] | 1.06 [-4.29 to 6.4]
Statistical Analysis 1: Comparison: Problem-Solving Treatment vs Supportive Psychotherapy; Test type: Superiority; cohen's d = .38

15. Other Pre Specified Outcome: Brief Pain Inventory (BPI)
Description: Brief Pain Inventory (BPI) measure of pain severity and interference. The total severity composite score ranges from 0-10 with higher scores indicating worse pain. The total pain interference score ranges from 0-10 with higher scores indicating more interference.
Time Frame: Change from Baseline to 12 weeks
Population: Only individuals who provided data were analyzed.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Problem-Solving Treatment | Supportive Psychotherapy
Number analyzed (Participants) | 19 | 13
score on a scale
  Composition | .33 [-.18 to .84] | -.13 [-.67 to .4]
  Interference | -.2 [-1.37 to .96] | .77 [-.13 to 1.67]
Statistical Analysis 1: Comparison: Problem-Solving Treatment vs Supportive Psychotherapy; Severity; Test type: Superiority; Cohens d = 0.47
Statistical Analysis 2: Comparison: Problem-Solving Treatment vs Supportive Psychotherapy; interference; Test type: Superiority; Cohens d = 0.46

16. Other Pre Specified Outcome: Brief Pain Inventory (BPI)
Description: as for outcome 15
Time Frame: Change from Baseline to 6 months
Population: Only individuals who provided data were analyzed.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Problem-Solving Treatment | Supportive Psychotherapy
Number analyzed (Participants) | 15 | 18
score on a scale
  Composite Score | .82 [-.04 to 1.68] | -.18 [-.95 to .59]
  Interference | .58 [-.81 to 1.97] | -.29 [-1.34 to .75]
Statistical Analysis 1: Comparison: Problem-Solving Treatment vs Supportive Psychotherapy; Severity Subscale; Test type: Superiority; Cohens d = 0.64
Statistical Analysis 2: Comparison: Problem-Solving Treatment vs Supportive Psychotherapy; Interference subscale; Test type: Superiority; Cohen's d = 0.38

ADVERSE EVENTS:
Time Frame: 6-months
Description: Adverse events were counts tabulated medical vs. psychiatric.
Arm/Group | Problem-Solving Treatment | Supportive Psychotherapy
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 4/22 | 2/22
Other Adverse Events (participants affected / at risk) | 21/22 | 15/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Problem-Solving Treatment (N=22) | Supportive Psychotherapy (N=22)
Increase in psychiatric symptoms (Psychiatric disorders) | 3 (3) | 2 (2)
Suspected transient ischemic attack (Cardiac disorders) | 1 (1) | 0 (0)
Increase in GI symptoms (Gastrointestinal disorders) | 1 (2) | 1 (1)
High blood sugar (Endocrine disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Problem-Solving Treatment (N=22) | Supportive Psychotherapy (N=22)
Psychiatric adverse event (Psychiatric disorders) | 3 (4) | 2 (2)
Medical adverse event (Investigations) | 19 (29) | 14 (37)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-30): https://cdn.clinicaltrials.gov/large-docs/65/NCT04490265/Prot_SAP_000.pdf
  • Informed Consent Form (2020-05-18): https://cdn.clinicaltrials.gov/large-docs/65/NCT04490265/ICF_001.pdf